CLINICAL TRIAL: NCT06896630
Title: Effect of Long-Term Use of Tenofovir (TDF) on Renal Function in Patients With Chronic Hepatitis B
Brief Title: Effect of Tenofovir (TDF) on Renal Function in Patients With Chronic Hepatitis B
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour shaaban Mohamed Abd elrasoul, Principal Investigator, Assiut University
Other Study IDs: TDF ON RENAL FUNCTION
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Tenofovir Disoproxil Fumarate; Renal Function Disorder; Chronic HBV Infection
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF) — ANTIVIRAL TREATMENT FOR CHRONIC HEPATITIS B VIRUS INFECTION

SUMMARY:
Effect of Long-Term Use of Tenofovir (TDF) on Renal Function in Patients with Chronic Hepatitis B Over a Five-Year Period

DETAILED DESCRIPTION:
Hepatitis B is a viral infection that affects 257 million people worldwide and approximately 820,000 die annually of HBV-related causes and is a leading cause of liver cirrhosis and hepato-cellular carcinoma . Thus, it is a global public health problem. The diagnosis of chronic hepatitis B (CHB) infection is based on the persistence of hepatitis B surface antigens (HBsAg) for more than six months . Some patients may experience acute exacerbation of the HBV infection and progression to acute-on chronic liver failure (ACLF), which has a high mortality rate in spite of substantial supporting and the use of a great quantity resources. Liver transplantation is a latent treatment election for most ACLF patients; hence, factors such as donor shortage and high cost restrict its clinical application.

Hence, Early intervention and treatment are very important in patients with ACLF.

The goals of antiviral therapy are to suppress viral replication and to ensure the loss of related antigens . Currently, there are two classes of antiviral drugs that are approved for the treatment of chronic Hepatitis B infection: Interferon alpha and Nucleoside analogues. Among the Nucleoside analogues, Entecavir (ETV), Tenofovir disoproxil fumarate (TDF), and Tenofovir alafenamide fumarate (TAF), are the most widely used as first-line treatments. The effectiveness of Nucleos(t)ide analogues (NUCs) is evident, and their usage is easier as they are administered orally and have fewer side effects. But most patients require long-term treatment as premature discontinuation of NUCs treatment may result in virological relapse and liver failure. TDF is one of the most potent antiviral agents against HBV and HIV. However, its potential effects on renal insufficiency are still being questioned . Tenofovir, Entecavir, and Telbivudine are more widely used due to their superior virological, biochemical, and clinical efficacy. They also have a higher barrier to resistance and more tolerable side effect profiles .The kidney is the primary route for the excretion of NUCs so that nephrotoxicity can be encountered during usage of these agents. Although the exact mechanism of nephrotoxicity is not well known, it can be attributed to alterations in renal tubular transporters especially in the proximal renal tubules, as well as apoptosis and mitochondrial toxicity. The tubular damage leads to defective proximal tubular secretion and reabsorption of several substances including phosphate, resulting in reduced serum phosphate levels, elevated phosphate levels in the urine and elevated serum levels of creatinine.

Tenofovir disoproxil fumarate (TDF), the prodrug of the Nucleotide analogue reverse transcriptase inhibitor (NRTI) Tenofovir, is active against both HIV and HBV. TDF use as part of antiretroviral therapy (ART) carries a risk of proximal tubular dysfunction and declining glomerular filtration rate (GFR), and monitoring of renal function is recommended during treatment . The risk is related to both level and length of TDF exposure and is enhanced by co-administration of pharmacological boosters (e.g., Ritonavir), low body weight, and pre-existing chronic kidney disease (CKD).

Whilst TDF discontinuation is generally associated with improved renal function, longer exposure and lower GFR at TDF interruption predict a reduced likelihood of GFR recovery.

ELIGIBILITY:
Inclusion Criteria:

Adult male or female patients aged 18 to 60 years.

Diagnosed as HBV-positive.

Long-term use of Tenofovir Disoproxil Fumarate (TDF) for more than five years.

Exclusion Criteria:

Presence of other chronic liver diseases.

Diagnosed with Chronic Kidney Disease (CKD), regardless of etiology.

Patients who refuse to participate in the study.

Patients on combination therapy, including:

Interferon and Nucleoside analogue combination therapy.

Multiple nucleoside analogue combination therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study Population Age Range: 18 to 60 years Sex: Male and Female HBV Status: HBV-positive patients Treatment Duration: Long-term use of Tenofovir (TDF) for more than five years Sampling Method: Non-Probability Sampling Healthy Volunteers: Not Accepted
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in eGFR in Patients on Long-Term Tenofovir (TDF) Therapy | BASELINE
  "Renal function will be assessed using estimated glomerular filtration rate (eGFR) calculated by the CKD-EPI equation
Assessment of Renal Function: Serum Creatinine in Patients on Long-Term Tenofovir (TDF) Therapy | BASELINE
  "Renal function will be assessed using serum creatinine levels measured through standard laboratory assays.
proteinuria will be evaluated through urine protein-to-creatinine ratio | BASELINE
  proteinuria will be evaluated through urine protein-to-creatinine ratio (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Effat AbdelHady Tony Ahmed, PROFESSOR OF NEPHROLOGY, Study Director — Assiut University; Mohamed Abdelhakim Omran Mahdy, LECTRURER, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liang RA, Hoiland II, Ueland T, Aukrust P, Snir O, Hindberg K, Braekkan SK, Garred P, Mollnes TE, Hansen JB. Plasma levels of mannose-binding lectin and future risk of venous thromboembolism. J Thromb Haemost. 2019 Oct;17(10):1661-1669. doi: 10.1111/jth.14539. Epub 2019 Jul 1. PMID 31220397
- [Background] Leggio M, Fusco A, D'Emidio S, Severi P, Lombardi M, Caldarone E, Armeni M, Mereu D, Bendini MG, Mazza A. Management of oral anticoagulation in patients with atrial fibrillation: newer agents, newer conundrums? J Intern Med. 2018 Dec;284(6):697-699. doi: 10.1111/joim.12755. Epub 2018 Apr 15. No abstract available. PMID 29658167
- [Background] Marques NDSF, Abreu LC, Santos BVD, Neto CFR, Silva JRCD, Braga KKS, Uchoa KDS, Moraes LMS, Ferreira LCP, Ribeiro NG, Santos SLD, Silva TAD, Andrade PE, Raimundo RD. Cardiorespiratory parameters and glycated hemoglobin of patients with type 2 diabetes after a rehabilitation program. Medicine (Baltimore). 2018 Feb;97(8):e9321. doi: 10.1097/MD.0000000000009321. PMID 29465549
- [Background] Alontseva DL, Ghassemieh E, Voinarovych S, Russakova A, Kyslytsia O, Polovetskyi Y, Toxanbayeva A. Characterisation of the microplasma spraying of biocompatible coating of titanium. J Microsc. 2020 Sep;279(3):148-157. doi: 10.1111/jmi.12849. Epub 2019 Dec 22. PMID 31797374
- [Background] Wang C, Chang D, Wang J, Gao Q, Zhang Y, Niu C, Liu C, Jia Y. Size and crystal symmetry breaking effects on negative thermal expansion in ScF3 nanostructures. Phys Chem Chem Phys. 2021 Nov 10;23(43):24814-24822. doi: 10.1039/d1cp02809j. PMID 34714310
- [Background] Tsai HJ, Chuang YW, Yang SS, Chang YZ, Chang HR, Lee TY. Evaluating the renal safety of tenofovir disoproxil fumarate in hepatitis B patients without chronic kidney disease. J Viral Hepat. 2021 Nov;28(11):1579-1586. doi: 10.1111/jvh.13603. Epub 2021 Sep 12. PMID 34464999